CLINICAL TRIAL: NCT04056039
Title: Efficacy of Atorvastatin vs Colchicine in Decrease of Troponin I of High Sensitivity as a Biomarker of Myocardial Damage in Patients With Rheumatoid Arthritis With Severe Activity.
Brief Title: Atorvastatin vs Colchicine in Decrease of Troponin I of High Sensitivity in Patients With Rheumatoid Arthritis.
Acronym: ACAR1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Responsible Party: Principal Investigator, José Alfredo Alvarado Alvarado, Internal Medicine Residency, Hospital Central "Dr. Ignacio Morones Prieto"
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AVSCAR001
Record Dates: First submitted 2019-06-21; First posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Cardiovascular Diseases; Arthritis, Rheumatoid
Keywords: rheumatoid arthritis; Troponin I; Atorvastatin; Colchicine; Cardiovascular disease risk
MeSH Terms: conditions — Cardiovascular Diseases; Arthritis, Rheumatoid | interventions — Atorvastatin; Colchicine

STUDY DESIGN:
Intervention Model Description: A pilot study with 30 patients per group, according to Browne, will be recalculated based on the preliminary result and the power of effect. This is a randomized controlled trial blind to the rheumatologist and the cardiologist who will carry out the evaluation of the patient. The randomization was performed in blocks. Description: Random assignment of n subjects with an equal number in all N conditions can be done by randomizing blocks, where the size of the block is the number of experimental conditions. The number of independent variables and the number of levels in each IV are specified as input. The output is a random design block.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "Atorvastatin" (Active Comparator): -Changes of troponin I in rheumatoid arthritis with "atorvastatin" 40 mg orally every 24 hours for four weeks
  Interventions: Drug: Atorvastatin
- "Colchicine" (Active Comparator): Changes of troponin I in rheumatoid arthritis with "colchicine" with an initial dose of 0.25 mg every 8 hours, with titration in the first 3 days according to tolerance up to a maximum dose of 0.5 mg every 8 hours for four weeks
  Interventions: Drug: Colchicine

INTERVENTIONS:
Drug: Atorvastatin — Efficacy of atorvastatin 40 mg orally every 24 hours for four weeks vs colchicine with an initial dose of 0.25 mg every 8 hours, with titration in the first 3 days according to tolerance up to a maximum dose of 0.5 mg every 8 hours for four weeks in decrease of troponin I of high sensitivity
  Arms: "Atorvastatin"
Drug: Colchicine — Efficacy of atorvastatin 40 mg orally every 24 hours for four weeks vs colchicine with an initial dose of 0.25 mg every 8 hours, with titration in the first 3 days according to tolerance up to a maximum dose of 0.5 mg every 8 hours for four weeks in decrease of troponin I of high sensitivity
  Arms: "Colchicine"

SUMMARY:
Pilot study. The primary end point is the evaluation the efficacy of treatment with atorvastatin compared to colchicine for the decrease of high sensitivity troponin I levels in patients with rheumatoid arthritis with severe activity according of the Disease Activity Score 28 (DAS 28> 5.1), through a randomized controlled clinical trial blinded to the rheumatologist and the cardiologist who will carry out the evaluation of the patient.

DETAILED DESCRIPTION:
A pilot study will be conducted in patients older than 18 years with a diagnosis of rheumatoid arthritis in the Hospital Central "Dr. Ignacio Morones Prieto", these patients will be evaluated by the rheumatologist and the patients with and patients with severe activity according of the Disease Activity Score 28 (DAS 28> 5.1) will be invited to their recruitment, a history of ischemic heart disease, heart failure or chronic kidney disease will be reviewed for its exclusion. This is a randomized controlled clinical trial blinded to the rheumatologist and the cardiologist who will carry out the evaluation of the patient. Patients who meet the aforementioned criteria, will be given informed consent to be signed, if accepted and signed, treatment will be given according to block randomization performed as follows: atorvastatin 40 mg orally every 24 hours for four weeks, colchicine with one initial dose of 0.25 mg every 8 hours titrating dose in the first 3 days according to tolerance up to 0.5 mg every 8 hours for four weeks.

A high-sensitivity troponin I measurement will be taken by means of a peripheral blood sample, the echocardiogram will be evaluated by the cardiologist, patients with heart failure will be eliminated with an unknown left ventricular ejection fraction or unknown ischemic heart disease and will be diagnosed at the first echocardiogram. We will review the laboratory studies of the evaluation with rheumatology: blood biometry, lipid profile, anti-citrullinated antibodies, rheumatoid factor, serum creatinine, uric acid, serum glucose. Patients from the area of rheumatology will be reviewed daily to recruit patients who meet the inclusion criteria, the patient will be informed in addition to signing the informed consent in case of accepting. The evaluation of the activity of the disease will be carried out using the DAS 28 scale at the beginning and end of the treatment. Follow up by telephone every week to patient for information of treatment follow-up and adverse effects. When reporting adverse effects with colchicine doses, the dose will be minimally tolerated or discontinued if necessary, as with treatment with atorvastatin. Peripheral blood samples for high sensitivity troponin I will be taken at the end of the four weeks, in addition to an echocardiogram in case of finding alterations in the first evaluation through this study. The changes in this cardiac biomarker and echocardiographic findings of said pilot study will be analyzed with the appropriate methods for this, their differences and statistical significance.

The primary end point is the evaluation the efficacy of treatment with atorvastatin compared to colchicine for the decrease of high sensitivity troponin I levels in patients with rheumatoid arthritis with severe activity (DAS 28> 5.1). Patients are randomized by means of a web-based procedure with a permuted-block design according to trial center. Patients are assigned in a 1:1 ratio to receive atorvastatin 40 mg orally every 24 hours for four weeks or colchicine with an initial dose of 0.25 mg every 8 hours, with titration in the first 3 days according to tolerance up to a maximum dose of 0.5 mg every 8 hours for four weeks.

Secondary end points are the evaluation of findings found in echocardiography in patients with rheumatoid arthritis with severe activity before and after treatment with atorvastatin or colchicine according to randomization and the evaluate the risk factors associated with a higher elevation high sensitivity troponin I in patients with rheumatoid arthritis.

Universe of study. Patients with rheumatoid arthritis older than 18 years with activity of the disease according to DAS 28> 5.1 attended in the rheumatology service of the Central Hospital "Dr. Ignacio Morones Prieto", San Luis Potosi, San Luis Potosi, Mexico.

Patients are eligible if they are older than 18 years with a diagnosis of rheumatoid arthritis according to the diagnostic criteria of the American College of Rheumatology and the European League against Rheumatism 2010 and severe activity by the scale of measurement of the disease (DAS) and sign the informed consent.

The exclusion criteria are patient with ischemic heart disease or heart failure with decreased left ventricular ejection fraction demonstrated by initial echocardiography, known chronic kidney disease and previous diagnosis of acute coronary syndrome or heart failure.

The elimination criteria are that the patient present an acute coronary syndrome requiring hospitalization or serious adverse effects in whom the suspension of treatment is necessary.

Variables in the study. Dependent variable. Levels of high sensitivity troponin I in ng / ml. Independent variable. Group 1 atorvastatin 40 mg orally every 24 hours for four weeks. Group 2 of colchicine with an initial dose of 0.25 mg every 8 hours, with titration in the first 3 days according to tolerance up to a maximum dose of 0.5 mg every 8 hours for four weeks.

Control variables. Age, Sex, Diabetes mellitus according to the diagnostic criteria of the American Diabetes Association, Hypertension according to the diagnostic criteria of the European Society of Hypertension and the European Society of Cardiology and Glomerular filtration rate.

The primary efficacy outcome was determined with the use of an unconditional logistic-regression model fitted to estimate.

STATISTIC ANALYSIS. The variables will be described by means of frequencies or percentages. The statistical analysis of each variable will be carried out with measures of central tendency and dispersion, the normality of the data will be evaluated. The variables with normal distribution will be expressed as mean and standard deviation. The qualitative data will be expressed as a percentage and frequency distribution. T student analysis of the means will be performed. A p less than 0.05 will be taken as statistical significance. All this will be done through the statistical program R version 3.4.3.

Sample's size calculation Initially, a pilot study with 30 patients per group, according to Browne, will be recalculated based on the preliminary result and the power of the effect.

This is an investigation with minimal risk. All the procedures will be in accordance with the stipulations of the Regulation of the General Law of Health in the Matter of Health Research. Title two, chapter I, Article 17, Section II.

Treatment and diagnostic maneuvers do not violate the rules of the Declaration of Helsinki adopted by the 18th World Medical Assembly, Helsinki, Finland, June 1964 and until amended at the 64th World Medical Assembly General Assembly, Fortaleza, Brazil, October 2013. To the Laws and Codes of Mexico such as Article 100 of the General Health Law and Article 20 where it states that consent by means of information is understood as the written agreement by which the subject of investigation, or where appropriate, your legal representative authorizes your participation in the investigation with full knowledge of the nature of the procedures and risks to which you will submit, with the ability to freely choose and without any coercion.

Patients who decide to collaborate in the study and who meet the selection criteria will be informed in writing what their participation will be and they will be asked to sign the informed consent form, being completely free to leave the project if so, they decide it, without this determining a decrease in the care of their medical attention. The information will be handled with strict confidentiality.

The study protocol was reviewed & approved by the ethical committee of the hospital Central "Dr. Ignacio Morones Prieto", with ethic number 63-18. Written knowledgeable consents were obtained from participants in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years with a diagnosis of rheumatoid arthritis according to the diagnoses of the American College of Rheumatology and the European League against rheumatism 2010 with severe disease activity according to DAS 28> 5.1.
* Patients who are accepted according to previous criteria and with signed informed consent.

Exclusion Criteria:

* Patients with a history of ischemic heart disease.
* Patients with a history of heart failure with decreased left ventricular ejection fraction
* Patients with chronic kidney disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Changes of high sensitivity troponin I levels | It will be evaluated before the start of treatment and at the end of the four weeks of treatment.
  Levels of high sensitivity troponin I in ng / ml with the ARCHITECT STAT Troponin-I assay of high sensitivity by immunoassay by chemo luminescent microparticles, with a calibration range of 0.0-50,000.00 pg / ml.

SECONDARY OUTCOMES:
Changes in echocardiographic findings | It will be evaluated before the start of treatment and at the end of the four weeks of treatment.
  Changes by echocardiography in patients with alterations found in the initial study after 4 weeks of treatment with a new imaging study.
Risk factors associated with a higher elevation high sensitivity troponin I | It will be evaluated before the start of treatment
  Perform statistical analysis with the baseline characteristics of patients to show their association with high levels of high sensitivity troponin I.

CONTACTS AND LOCATIONS:
Overall Officials: Juan M Lopez, MD, Study Chair — Ethics committee of the Hospital Central "Dr Ignacio Morones Prieto"; Emmanuel Rivera, MD, Study Chair — Research committee of the Hospital Central "Dr Ignacio Morones Prieto"
Locations (1):
- Hospital Central "Dr Ignacio Morones Prieto", San Luis Potosí City, Mexico

REFERENCES:
- [Background] Smolen JS, Aletaha D, Barton A, Burmester GR, Emery P, Firestein GS, Kavanaugh A, McInnes IB, Solomon DH, Strand V, Yamamoto K. Rheumatoid arthritis. Nat Rev Dis Primers. 2018 Feb 8;4:18001. doi: 10.1038/nrdp.2018.1. PMID 29417936
- [Background] Kitas G, Banks MJ, Bacon PA. Cardiac involvement in rheumatoid disease. Clin Med (Lond). 2001 Jan-Feb;1(1):18-21. doi: 10.7861/clinmedicine.1-1-18. No abstract available. PMID 11358070
- [Background] Gabriel SE. Cardiovascular morbidity and mortality in rheumatoid arthritis. Am J Med. 2008 Oct;121(10 Suppl 1):S9-14. doi: 10.1016/j.amjmed.2008.06.011. PMID 18926169
- [Background] Crowson CS, Liao KP, Davis JM 3rd, Solomon DH, Matteson EL, Knutson KL, Hlatky MA, Gabriel SE. Rheumatoid arthritis and cardiovascular disease. Am Heart J. 2013 Oct;166(4):622-628.e1. doi: 10.1016/j.ahj.2013.07.010. Epub 2013 Aug 29. PMID 24093840
- [Background] Khalid U, Egeberg A, Ahlehoff O, Lane D, Gislason GH, Lip GYH, Hansen PR. Incident Heart Failure in Patients With Rheumatoid Arthritis: A Nationwide Cohort Study. J Am Heart Assoc. 2018 Jan 19;7(2):e007227. doi: 10.1161/JAHA.117.007227. PMID 29352092
- [Background] Liao KP, Solomon DH. Traditional cardiovascular risk factors, inflammation and cardiovascular risk in rheumatoid arthritis. Rheumatology (Oxford). 2013 Jan;52(1):45-52. doi: 10.1093/rheumatology/kes243. Epub 2012 Sep 16. PMID 22986289
- [Background] Prasad M, Hermann J, Gabriel SE, Weyand CM, Mulvagh S, Mankad R, Oh JK, Matteson EL, Lerman A. Cardiorheumatology: cardiac involvement in systemic rheumatic disease. Nat Rev Cardiol. 2015 Mar;12(3):168-76. doi: 10.1038/nrcardio.2014.206. Epub 2014 Dec 23. PMID 25533796
- [Background] Karpouzas GA, Estis J, Rezaeian P, Todd J, Budoff MJ. High-sensitivity cardiac troponin I is a biomarker for occult coronary plaque burden and cardiovascular events in patients with rheumatoid arthritis. Rheumatology (Oxford). 2018 Jun 1;57(6):1080-1088. doi: 10.1093/rheumatology/key057. PMID 29554376
- [Background] de Boer RA, Nayor M, deFilippi CR, Enserro D, Bhambhani V, Kizer JR, Blaha MJ, Brouwers FP, Cushman M, Lima JAC, Bahrami H, van der Harst P, Wang TJ, Gansevoort RT, Fox CS, Gaggin HK, Kop WJ, Liu K, Vasan RS, Psaty BM, Lee DS, Hillege HL, Bartz TM, Benjamin EJ, Chan C, Allison M, Gardin JM, Januzzi JL Jr, Shah SJ, Levy D, Herrington DM, Larson MG, van Gilst WH, Gottdiener JS, Bertoni AG, Ho JE. Association of Cardiovascular Biomarkers With Incident Heart Failure With Preserved and Reduced Ejection Fraction. JAMA Cardiol. 2018 Mar 1;3(3):215-224. doi: 10.1001/jamacardio.2017.4987. PMID 29322198
- [Background] Divard G, Abbas R, Chenevier-Gobeaux C, Chanson N, Escoubet B, Chauveheid MP, Dossier A, Papo T, Dehoux M, Sacre K. High-sensitivity cardiac troponin T is a biomarker for atherosclerosis in systemic lupus erythematous patients: a cross-sectional controlled study. Arthritis Res Ther. 2017 Jun 13;19(1):132. doi: 10.1186/s13075-017-1352-7. PMID 28610589
- [Background] Evans JDW, Dobbin SJH, Pettit SJ, Di Angelantonio E, Willeit P. High-Sensitivity Cardiac Troponin and New-Onset Heart Failure: A Systematic Review and Meta-Analysis of 67,063 Patients With 4,165 Incident Heart Failure Events. JACC Heart Fail. 2018 Mar;6(3):187-197. doi: 10.1016/j.jchf.2017.11.003. Epub 2018 Jan 10. PMID 29331272
- [Background] Papageorgiou N, Briasoulis A, Lazaros G, Imazio M, Tousoulis D. Colchicine for prevention and treatment of cardiac diseases: A meta-analysis. Cardiovasc Ther. 2017 Feb;35(1):10-18. doi: 10.1111/1755-5922.12226. PMID 27580061
- [Background] Nidorf SM, Eikelboom JW, Budgeon CA, Thompson PL. Low-dose colchicine for secondary prevention of cardiovascular disease. J Am Coll Cardiol. 2013 Jan 29;61(4):404-410. doi: 10.1016/j.jacc.2012.10.027. Epub 2012 Dec 19. PMID 23265346
- [Background] Deftereos S, Giannopoulos G, Panagopoulou V, Bouras G, Raisakis K, Kossyvakis C, Karageorgiou S, Papadimitriou C, Vastaki M, Kaoukis A, Angelidis C, Pagoni S, Pyrgakis V, Alexopoulos D, Manolis AS, Stefanadis C, Cleman MW. Anti-inflammatory treatment with colchicine in stable chronic heart failure: a prospective, randomized study. JACC Heart Fail. 2014 Apr;2(2):131-7. doi: 10.1016/j.jchf.2013.11.006. PMID 24720919
- [Background] Li GM, Zhao J, Li B, Zhang XF, Ma JX, Ma XL, Liu J. The anti-inflammatory effects of statins on patients with rheumatoid arthritis: A systemic review and meta-analysis of 15 randomized controlled trials. Autoimmun Rev. 2018 Mar;17(3):215-225. doi: 10.1016/j.autrev.2017.10.013. Epub 2018 Jan 31. PMID 29353098
- [Background] Alvarado Cardenas M, Marin Sanchez A, Lima Ruiz J; en representacion del Grupo para estudio de Autoinmunidad y Estatinas. [Statins and autoimmunity]. Med Clin (Barc). 2015 Nov 6;145(9):399-403. doi: 10.1016/j.medcli.2014.11.017. Epub 2015 Feb 7. Spanish. PMID 25662717
- [Background] Fatemi A, Moosavi M, Sayedbonakdar Z, Farajzadegan Z, Kazemi M, Smiley A. Atorvastatin effect on systemic lupus erythematosus disease activity: a double-blind randomized clinical trial. Clin Rheumatol. 2014 Sep;33(9):1273-8. doi: 10.1007/s10067-014-2654-7. Epub 2014 May 13. PMID 24820145
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- [Background] Friede T, Kieser M. Sample size recalculation in internal pilot study designs: a review. Biom J. 2006 Aug;48(4):537-55. doi: 10.1002/bimj.200510238. PMID 16972704
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. Pilot Feasibility Stud. 2016 Oct 21;2:64. doi: 10.1186/s40814-016-0105-8. eCollection 2016. PMID 27965879

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/39/NCT04056039/SAP_000.pdf
  • Informed Consent Form (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/39/NCT04056039/ICF_001.pdf